CLINICAL TRIAL: NCT03318965
Title: Combination of APACHE Scoring Systems With Adductor Pollicis Muscle Thickness for the Prediction of Mortality in ICU
Brief Title: Scoring Systems in ICU and Malnutrition
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Other Study IDs: 1374103
Record Dates: First submitted 2017-10-10; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Critical Illness
Keywords: Mortality; Anthropometry; Nutrition Assessment; Caliper
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the present study was to compare the ability of acute physiology and chronic health evaluation (APACHE) scoring systems with the combination of an anthropometric variable score "adductor pollicis muscle (APM) thickness" to the APACHE systems in predicting mortality in the ICU. Three hundred and four patients enrolled in this prospective observational study. The APM thickness in dominant hand and APACHE II and III scores were measured for each patient upon admission. Given scores for the APM thickness, were added to APACHE score systems to make two composite scores of APACHE II- APM and APACHE III- APM. The accuracy of the two composite models and APACHE II and III systems in predicting mortality of patients was compared using area under the ROC curve.

Based on the study results, the area under the ROC curves improved in composite models. Therefore, it seemed that considering anthropometric variables may improve prediction of mortality in APACHE systems.

DETAILED DESCRIPTION:
The baseline medical history, physical examination, Acute Physiology and Chronic Health Evaluation score II and III (APACHE) were recorded for all patients. All data were collected by a single physician. The APACHE II and III scores were gathered using the method presented by Knaus. The dominant hand APM thickness (as reported by the patient, or the relative) was assessed by Caliper (Vogel, Germany) in the emergency room or at the time of the ICU admission. To estimate weight for the APM thickness, multivariate logistic regression analysis was used to determine the relation between mortality and the APM thickness while controlling for other physiologic variables (12 physiologic variables for APACHE II and 18 physiologic variables for APACHE III).The area under the receiver-operating curves (ROC curve) to predict mortality was used to compare APACHE II, APACHE III, APACHE II- APM and APACHE III- APM systems.

ELIGIBILITY:
Inclusion Criteria:

* Older than 16 years of age

Exclusion Criteria:

* Splints, in the upper extremities
* Casts in the upper extremities
* Edema in the upper extremities
* Patients with readmission during the study period
* Those transferred from other ICUs

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 304 eligible critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Prediction of Mortality | First day of ICU admission
  Mortality prediction by APACHE -APM

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, PhD, Study Chair — Shahid Beheshti University